CLINICAL TRIAL: NCT02022072
Title: Measurement of Assisted Vital Capacity to Appreciate the Level of Recruitment in Neuromuscular Diseases
Brief Title: Evaluation of Vital Capacity
Acronym: CVassist
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: With 50 patients, the measure of assist vital capacity has been validated
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-A00218-37
Record Dates: First submitted 2013-11-05; First posted 2013-12-27 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Respiration Disorders; Neuromuscular Disease
MeSH Terms: conditions — Respiration Disorders; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- measure of assisted vital capacity by mechanical insufflation (Other): measure of assisted vital capacity by a mechanical insufflation/exsufflation
  Interventions: Device: measures of assisted vital capacity by a mechanical insufflation/exsufflation (Cough Assist®)

INTERVENTIONS:
Device: measures of assisted vital capacity by a mechanical insufflation/exsufflation (Cough Assist®) — measures of assisted vital capacity by a mechanical insufflation/exsufflation (Cough Assist®)

SUMMARY:
Respiratory failure is the most common cause of death in neuromuscular diseases. The aim of this research is to evaluate the thoracopulmonary recruitment by comparison of inspiratory vital capacity (VC ins)and inspiratory/expiratory vital capacity (VC ins-ex) with the vital capacity (VC) according to pathology and severity of pulmonary damage of patients with neuromuscular diseases. The methodology consists in realize VC by support of inspiratory/expiratory pressures, while the patient is passive and realizing a maximal inspiratory/expiratory effort simultaneously, with the aid of mechanical insufflation/exsufflation device (Cough Assist®). The evaluation will last for 30 minutes and the non-inclusion criteria are those for an insufflation. The study hypothesis is that long term insufflation/exsufflation device use could improve thoracopulmonary mobility.

ELIGIBILITY:
Inclusion Criteria:

* consent form signature
* Men and women aged over or equal to 18 years old
* Medical examination before the research
* Negative results of tests of pregnancy for the women at age to procreate or taking an effective contraceptive
* Patients with neuromuscular pathologies without tracheostmy - Vital Capacity < 80% of theoretical value

Exclusion Criteria:

* Refuse to participate at the research
* Patient under guardianship or under trusteeship
* pregnant Women
* Patients unable to cooperate
* Patients without a security social scheme (as beneficiary or bearer of rights)
* Usual contra-indications for an insufflation (haemoptise, recent pneumothorax, pulmonary emphysema, pleuresy, nausea, chronic obstructive pulmonary diseasee or asthma, recent lobectomy, intracranial hypertension, troubles of consciousness, unable to talk)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Difference between spontaneous vital capacity and supported vital capacity at the inspiration and at inspiration/expiration at the same manoeuver. | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital R Poincare, Garches, France